CLINICAL TRIAL: NCT04621656
Title: Sugar Challenge Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: January, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1280111
Record Dates: First submitted 2020-10-30; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Type 2 Diabetes; Pre-Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Biospecimen Retention: Samples With DNA — Stool samples optimized for Microbiome and Functional Microbial studies. Blood, urine, saliva and/or buccal swabs for potential laboratory testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type 2 Diabetes: Individuals that have been previously diagnosed with Type 2 Diabetes. Those with Fasting Blood Glucose levels 126 mg/dL in two separate tests and/or HbA1C values greater than 6.5%. Individuals may take Metformin, SGLT2 inhibitors, of GLP-1 therapeutics. Not including those using Insulin therapeutics.
  Interventions: Combination Product: January Mobile Application (Sugar AI)
- Pre-Diabetes: Individuals that have been previously diagnosed with Pre-Diabetes. This group may include individuals with pre-diabetes that may be unaware of their condition. HbA1C values between 5.7% and 6.4%.
  Interventions: Combination Product: January Mobile Application (Sugar AI)
- Healthy: Individuals that have not been previously diagnosed with Metabolic Syndromes including Type 2 Diabetes, obesity, or increased levels of blood sugar. HbA1C values below 5.7%.
  Interventions: Combination Product: January Mobile Application (Sugar AI)

INTERVENTIONS:
Combination Product: January Mobile Application (Sugar AI) — Sugar AI is a mobile health and fitness app the allows participants to log and record health-related data through Continuous Glucose Monitors, Heart Rate Monitors, and manual food, water, and activity logging. Using machine learning data science techniques, the Sugar AI App integrates the data collected to personalize lifestyle recommendations and help individuals optimize their health and wellness.

SUMMARY:
This is a longitudinal study involving use of the January App which collects multiple data streams and employs machine learning techniques to offer personalized lifestyle recommendations and structured food and activity challenges.

DETAILED DESCRIPTION:
The Sugar Challenge Study is a real-world, longitudinal study aimed at understanding the impact of lifestyle (i.e. food choices, physical activity and sleep patterns), genetics and personalized lifestyle recommendations on blood glucose levels, blood pressure, immune system status, stress hormone levels and microbiome composition. The purpose of this 10-day observational study was to primarily elucidate the impact of food choices, physical activity, and sleep patterns on an individual's blood glucose. In addition, we probed if continuous and personalized feedback to participants would improve glycemic control acutely through better decision making. Multiple investigations may be performed over an indefinite period of time to improve the understanding of these interconnected relationships. For example, we will perform studies to understand an individual's blood glucose response to an oral glucose load or mixed meal. We will also perform studies to determine the phenotype (clinical, metabolic, or immunologic) associated with a particular genotype. The data collected will be analyzed using proprietary machine learning methods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, have pre-diabetes or metabolic syndrome or type 2 diabetes on metformin or GLP-1 or SGLT-2 therapy
* Have access to smart-phone with NFC reader
* Be willing to wear a continuous glucose monitor (CGM) and a smartwatch 24 hours/day for 10-14 consecutive days at a time
* Be willing to limit swimming to a maximum of 30 minutes per session while wearing CGM
* Available for two in-person or remote study visits (study orientation and close-out)
* Willing to provide weight at baseline and comprehensive logging of their activity, food and water consumption for 10-14 days
* Covered by health insurance plan
* Able and willing to give informed consent for study participation

Exclusion Criteria:

* Use of vitamin C supplements in excess of 200% of the United States Recommended Daily Allowance at least 14 days prior to starting the trial
* Allergy to skin adhesives used in the trial
* Women who are pregnant, lactating, have given birth in the past 6 months, or are planning to get pregnant in the next 6 months
* Individuals deemed unfit for participation by study physician
* Allergy to nuts
* Individuals who are taking any of the following medications:
* Insulin
* Progesterone
* Atypical antipsychotics
* Oral or injectable antidiabetic medications EXCEPT for metformin or Glucagon-like peptide-1 (GLP-1) agonists or Selective sodium-glucose transporter-2 (SGLT-2) inhibitors
* Oral corticosteroid use
* Triphasic oral contraceptives
* Blood thinners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals that volunteer for study through web-based advertisement. Includes predefined sub-populations of healthy individuals, pre-diabetes, and Type 2 Diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 1022 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of percent of total time monitored that blood glucose is in range 70-180 mg/dL | 10 Continuous Days
  The percentage of time an individual remains within a target blood glucose range through the measure of Continuous Glucose Monitor. Ranges defined by the American Diabetes Association (ADA). Current guidelines in range are to 70% of time within 70-180 mg/dL range.

SECONDARY OUTCOMES:
Assessment of change in the mean daily fasting glucose | 10 days
Assessment of change in the mean daily postprandial glucose levels | 10 days
Assessment of change in the mean daily total caloric intake | 10 days
Assessment of change in the daily number of meals consumed | 10 days
Assessment of micro and macronutrients of meals consumed through manual food logging. | 10 days
  Participants will log foods using a proprietary food database consisting of 18M+ items
Assessment of change in the daily caloric composition of meals consumed through manual food logging. | 10 days
  Composition will be calculated based on a cross reference of the logged meal with a proprietary food database to yield caloric contributions of each food item.
Assessment of change in physical activity as measured by heart rate monitor coupled to participant logs. | 10 days
Assessment of change in sleep quality and pattern as measured by heart rate monitor coupled to participant logs. | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- January, Inc., Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: Yes
To inform participant and primary care physician of abnormal CGM levels.
Supporting Information: CSR
Time Frame: 30 Days following 10 day participation
Access Criteria: Reporting a notification of abnormal CGM data to participant. Primary care physician has access to CGM glucose values on request.